CLINICAL TRIAL: NCT00269178
Title: Cluster Randomized Trial of the Impact of a Peer-health Education Programme on Malaria Knowledge Attitudes and Practice in Students and Their Families
Brief Title: Cluster Randomized Trial of Peer Health Education in Malaria in The Gambia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Medical Research Council Unit, The Gambia (Other); Nova Scotia Gambia Association, The Gambia (Unknown); Centre for Innovation Against Malaria, The Gambia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SCC L2002.69; SSC L2002.69
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2024-11-26 (Actual); Status verified 2003-03

CONDITIONS: Malaria
Keywords: malaria; knowledge attitudes and practice (KAP); bednets; peer health education
MeSH Terms: conditions — Malaria

INTERVENTIONS:
Behavioral: Peer Health Education Programme

SUMMARY:
Health promotion in schools aims to improve the health and well being of students by empowering them with the knowledge, skills and confidence to take responsibility for their own health. We incorporated a malaria component to an established peer health education programme in schools in The Gambia, and evaluated its impact on knowledge attitudes and practice (KAP) of school students and their families using a cluster randomized design. Since malaria is a particular problem among children under 5 and pregnant women, students were encouraged to explain what they learned to their families, and we sought to evaluate whether the malaria messages were taken up by the students' families. Evaluation endpoints are KAP in students, and KAP in women living in the school students' home compound.

DETAILED DESCRIPTION:
12 communities in The Gambia, each including an upper basic and/or a senior secondary school, were pair-matched on urban/rural location and school type, and one community in each pair randomly selected to receive the peer-health education programme immediately or after a delay, to permit evaluation. The intervention programme comprised training of peer health educators, teacher coordinators, and members of drama troupes, in key malaria messages and principles of health education. The peer educators then conducted a rolling programme of presentations to children and youth in their own schools using drama, puppetry, small group and in-class presentations about malaria, as well as community outreach programs targeting out-of-school youth and the general public. In each school a systematic sample of 75 students were interviewed 10 weeks and 6 months after the start of the programme, and in each school catchment area a sample of 80 women were interviewed at the same time, and bednet use by children under 5 yrs in their care was recorded. From the interviews scores were derived for knowledge about malaria treatment and prevention and knowledge scores and net coverage in children compared between intervention and control schools.

ELIGIBILITY:
Inclusion Criteria:

* Woman caring for a child under 5 years of age, living in the compound of one of the peer health educators
* Student attending school

Exclusion Criteria:

* Not caring for a child under 5 years (for women)
* Not living in a compound of a peer health educator (for women)

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 960
Dates: Start 2003-08; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
1. Bednet use among children under 5yrs of age living in the household of peer health educators 10 wweks and 6 months after the start of the intervention
2. Malaria knowledge attitudes and practice among women in the family of peer health educators 10 week and 6 months after the start of the intervention
3. Malaria knowledge attitudes and practice among school students 10 weeks and 6 months after the start of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Paul JM Milligan, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Medical Research Council Laboratories, Banjul, The Gambia